CLINICAL TRIAL: NCT04654936
Title: Feasibility and Acceptability of a 12 Week Online Dietary Intervention Promoting the MIND Diet Using the COM-B Model
Brief Title: Effectiveness of a 12 Week Theory Driven Intervention Promoting Adherence to the MIND Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Responsible Party: Principal Investigator, Deirdre Timlin, Principle investigator, University of Ulster
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: DTimlin
Record Dates: First submitted 2020-11-05; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Cognitive Change

STUDY DESIGN:
Intervention Model Description: This study includes 2 intervention arms and one control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MIND diet with support (Experimental): This intervention group are to follow the MIND diet guidelines for 12 weeks with the support of a 12 week online theory driven website and resources
  Interventions: Behavioral: MIND diet
- MIND diet no support (Experimental): This group are to follow the MIND diet guidelines with no website support
  Interventions: Behavioral: MIND diet with no support
- Control (No Intervention): The group follow usual diet

INTERVENTIONS:
Behavioral: MIND diet — 12 week MIND diet study: Participants access a website that is theory driven using the Behaviour Change Wheel to help motivate and promote MIND diet adherence. Participants are to consume MIND diet foods daily and meet MIND diet weekly recommendations
  Arms: MIND diet with support
Behavioral: MIND diet with no support — Participants are to consume MIND diet food recommendations over a 12 week period with no support except for a self-monitoring resource and MIND diet guidelines
  Arms: MIND diet no support

SUMMARY:
This study aims to test the feasibility and acceptability of a 12 week online dietary promoting MIND diet behaviour. This study also tests the effectiveness of the MIND diet on cognitive function, mood, quality of life and participants capability, opportunity and motivation towards adoption of the MIND diet.

DETAILED DESCRIPTION:
This study is a randomized controlled prospective follow up study, condition (control Vs intervention) x time(baseline Vs follow up) ANOVA with repeated measures design. Outcome measures for COM-B, cognitive function, mood and quality of life were recorded for both the intervention and control groups. With power set at .80, and alpha = .05, G*Power indicated that a sample size of 36 would be required. Forty-one participants took part in the study. Participants were healthy male, and female aged between 40-55 years old living in Northern Ireland.

There are 2 intervention arms and one control group. The intervention was designed using the Behaviour Change Wheel, with prior qualitative research informing the intervention.

All statistical analyses were performed using the Statistical Package for the Social Sciences (SPSS) with significance set at P < 0.05 throughout

ELIGIBILITY:
Inclusion Criteria:

. Healthy male and female aged 40-55 living in NI

Exclusion Criteria:

* Anyone on a specific dietary pattern (veganism, vegetarian, Atkins)
* Anyone on a specific diet recommended by their Doctor (eating disorder)
* Specific illnesses such as high cholesterol, diabetes, heart disease, dementia.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-11-06 (Actual)

PRIMARY OUTCOMES:
Cognitive function | 12 weeks
  Tests used for this study were spatial working memory (SWM), spatial span (SSP), pattern recognition memory (PRM) and reaction time (RTI). These tests are computerised and measure the length of time it takes to complete task in milliseconds.

SECONDARY OUTCOMES:
Mood | 12 weeks
  Positive and Negative Affect Scale bref was used to measure mood 4 times a day over 4 days at baseline and follow-up. The maximum score for positive affect is 50 with higher scores representing higher levels of positive affect. Negative affect scores are a maximum of 50 with lower scores representing lower levels of negative affect.
World Health Organisation Bref Quality of life | 12 weeks
  WHO bref questionnaire was used to measure quality of life at baseline and follow up. The maximum score is 100, with higher scores representing higher quality of life.
Capability, opportunity, motivation and behaviour model | 12 weeks
  COM-B questionnaire measuring participants capability opportunity and motivation towards adoption of the MIND diet at baseline and follow up. Maximum scores are 110 with higher scores representing higher capability, opportunity, motivation towards MIND diet behaviour.

CONTACTS AND LOCATIONS:
Overall Officials: Liz Simpson, PhD, Principal Investigator — Ulster University
Locations (1):
- Life and Health Science, Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Timlin D, McCormack JM, Kerr M, Keaver L, Simpson EEA. The MIND diet, cognitive function, and well-being among healthy adults at midlife: a randomised feasibility trial. BMC Nutr. 2025 Mar 25;11(1):59. doi: 10.1186/s40795-025-01020-6. PMID 40134050